CLINICAL TRIAL: NCT02334709
Title: Phase I/II Trial of Stereotactic Body Radiotherapy With Concurrent Fixed Dose Tyrosine Kinase Inhibitors in Metastatic Renal Cell Carcinoma: Dose Limiting Toxicity and Abscopal Effect.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Radiotherapie, Study Principal Investigator, University Hospital, Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2013/1087
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiosurgery

ARMS (1):
- SBRT + fixed dose Tyrosine Kinase Inhibitor (Experimental): Single arm phase I trial with 3 dose-escalation arms
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — A first line TKI will be administered according to the standard dosing of the drug for metastatic RCC during a 1-week run-in period after which SBRT will be delivered to the largest metastatic lesion concurrently with the TKI. The SBRT dose will be escalated in 3 dose levels, starting at 24Gy (8 Gy per fraction), followed by 30 Gy (10 Gy per fraction) and 36 Gy (12 Gy per fraction).

SUMMARY:
Tyrosine kinase inhibitors (TKIs) are often used in the standard treatment for patients with metastasized renal cell carcinoma. In addition to their ability to specifically inhibit tumor growth, TKIs also interfere with the vascularisation of the tumor. Unfortunately, most patients do not obtain long-lasting clinical benefit from this treatment. The goal of the current study is to enhance the effect of TKIs by combining them with stereotactic radiotherapy treatment of one of the metastases. This type of radiotherapy allows us to precisely irradiate the tumor with minimal effect on the surrounding healthy tissue. Recently it has been demonstrated that this type of radiotherapy stimulates the immune system to attack the tumor. By combining stereotactic radiotherapy with TKIs we expect to observe a reduction of metastases in a bigger population of patients.

In the first part of our study we focus on the safety of the combination therapy. In the second part we will evaluate the combined treatment response.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* diagnosis of RCC with clear-cell component histology
* at least 3 extracranial measurable metastatic lesions per RECIST
* Karnofsky Performance score >60
* patients should have undergone cytoreductive treatment of their RCC at least 6 weeks prior to inclusion
* patients should have adequate organ function for TKI treatment.

Exclusion Criteria:

* prior systemic treatment for RCC
* uncontrolled central nervous metastases
* prior radiotherapy interfering with SBRT
* any disorder precluding understanding of trial information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 2 years
  Dose limiting toxicity will be assessed before start of TKI, before SBRT, at the end of SBRT and at each follow-up visit

SECONDARY OUTCOMES:
Response rate | 4 years
  Response rate will be evaluated at 12 weeks following the start of TKI.
Immunomonitoring | 4 years
  Immunomonitoring before start of TKI, before SBRT and 2 weeks after SBRT.

CONTACTS AND LOCATIONS:
Overall Officials: Piet Ost, PhD, Principal Investigator — Dept. of Radiotherapy, Ghent University Hospital
Locations (1):
- Dept. of Radiotherapy, Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

REFERENCES:
- [Derived] De Wolf K, Rottey S, Vermaelen K, Decaestecker K, Sundahl N, De Lobel L, Goetghebeur E, De Meerleer G, Lumen N, Fonteyne V, De Maeseneer D, Ost P. Combined high dose radiation and pazopanib in metastatic renal cell carcinoma: a phase I dose escalation trial. Radiat Oncol. 2017 Sep 22;12(1):157. doi: 10.1186/s13014-017-0893-x. PMID 28938918